CLINICAL TRIAL: NCT04555486
Title: A Phase 1 Placebo-Controlled, Double-Blind, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Dose of DCR-PHXC in Patients With Primary Hyperoxaluria Type 3
Brief Title: Study to Evaluate Safety, Tolerability, PK and PD of DCR-PHXC in PH Type 3 Patients
Acronym: PHYOX4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCR-PHXC-104
Record Dates: First submitted 2020-09-02; First posted 2020-09-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary Hyperoxaluria Type 3
Keywords: primary hyperoxaluria; primary hyperoxaluria type 3; primary hyperoxaluria 3; PH; PH type 3; PH3; RNAi; RNAi therapeutic; LDHA; LDH; GalNAc; siRNA; nedosiran; DCR-PHXC
MeSH Terms: conditions — Hyperoxaluria, Primary | interventions — nedosiran

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two interventions: the study drug DCR-PHXC (also known as nedosiran) or the placebo comparator Sterile Normal Saline. For every 2 participants that receive DCR-PHXC, 1 participant will receive placebo. Thus, 4 participants are expected to receive DCR-PHXC, and 2 participants are expected to receive placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DCR-PHXC (Experimental): Participants that are at least 12 years old will receive a single dose of 3 mg/kg DCR-PHXC (or nedosiran) via subcutaneous (SC) injection. Participants that are 6-11 years old will receive a single dose of 3.5 mg/kg DCR-PHXC (nedosiran) via SC injection.
  Interventions: Drug: DCR-PHXC
- Sterile Normal Saline (0.9% NaCl) (Placebo Comparator): Participants will receive a single dose of Sterile Normal Saline (0.9% NaCl) for subcutaneous (SC) injection, administered at same injection volume as DCR-PHXC, to serve as placebo.
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: DCR-PHXC — Intervention, drug, DCR-PHXC
  Other Names: Nedosiran
  Arms: DCR-PHXC
Drug: Sterile Normal Saline (0.9% NaCl) — Placebo comparator
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The DCR-PHXC-104 study is designed to assess the safety, tolerability, and pharmacological parameters of a single dose of DCR-PHXC in Primary Hyperoxaluria Type 3 (PH3). Participants should have had at least one stone event within 12 months of screening and intact renal function.

DETAILED DESCRIPTION:
Potential participants are screened over an up-to-35-day period (with an extra 7-day period for participants who are required to repeat screening 24-hour urine collections or initially unanalyzable screening laboratory assessment samples) prior to randomization. Eligible participants will receive a single dose of DCR-PHXC or placebo on Day 1.

In order to maintain the treatment blind, 24-hour urine oxalate (Uox) results that could unblind the study will not be reported to investigative sites or other blinded personnel until the study has been unblinded.

It is expected that approximately 10 participants will be screened in order to randomize 6 participants (2:1 randomization; 4 nedosiran:2 placebo) to the study.

Following the up-to-6-week screening period, participants will return to the clinic for interim visits up to Day 85. Visits occurring between the Day 1 and the Day 85 visit may be conducted as at-home telemedicine visits at the discretion of the Investigator. The total time on study for each participant is approximately 18 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Genetically confirmed PH3
* 24-hour Uox excretion ≥ 0.7 mmol (adjusted per 1.73 m^2 body surface area [BSA] in participants < 18 years of age) on both assessments conducted in the screening period
* Less than 20% variation between the two 24-hour urinary creatinine excretion values (mmol/kg/24 hours) in the screening period
* Estimated glomerular filtration rate (eGFR) at screening ≥ 30 mL/min, normalized to 1.73 m^2 BSA
* History of at least one stone event within the last 12 months. Stone events are defined as any of the following:

  * renal stone requiring medical intervention, e.g., outpatient procedures such as lithotripsy, or hospitalization or inpatient surgical intervention for confirmed stone-related pain and/or complications;
  * stone passage with or without hematuria; or
  * renal colic requiring medication.

Key Exclusion Criteria:

* Documented evidence of clinical manifestations of systemic oxalosis (including pre-existing retinal, heart, or skin calcifications, or history of severe bone pain, pathological fractures, or bone deformations)
* Plasma oxalate > 30 μmol/L

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Safety profile of a single dose of DCR-PHXC in PH3 Patients | Screening through Day 85
  Number of patients with abnormalities in clinically significant laboratory results, vital signs, and 12-lead ECG findings

SECONDARY OUTCOMES:
Plasma pharmacokinetics (PK) of a single dose of DCR-PHXC in PH3 patients | Day 1 (dosing) through Day 29
  Measure maximum plasma concentration of DCR-PHXC
The proportion of participants achieving a > 30% decrease from baseline in 24-hour Urine Oxalate (Uox) on 2 consecutive visits | After screening, 24-hour Uox will be measured at Days 29, 43, 57, and 85.
  Participants must maintain at least a 30% decrease from the average of 2 screening 24-hour Uox values to be considered "responders" to treatment. The proportion of responders to non-responders will be utilize to assess the efficacy of a single dose of DCR-PHXC in PH3 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Haagensen, MD, MBA, Study Director — Dicerna Pharmaceuticals
Locations (6):
- United States (3):
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, New York, New York
- Clinical Trial Site, Bonn, Germany
- Clinical Trial Site, Amsterdam, Netherlands
- Clinical Trial Site, London, United Kingdom